CLINICAL TRIAL: NCT03897309
Title: A Ph 1b, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Safety and Immunogenicity Study of Adenoviral-vector Based Oral Norovirus Vaccines Expressing GI.1 or GII.4 VP1 With Monovalent or Bivalent Dosing
Brief Title: Safety & Immunogenicity Study of Ad5 Based Oral Norovirus Vaccines
Acronym: VXA-NVV-103
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VXA-NVV-103
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Norovirus Infection
MeSH Terms: conditions — Caliciviridae Infections

STUDY DESIGN:
Intervention Model Description: Open-label sentinel followed by Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study subjects, study site and study team will remain blinded to treatment during study period 1 (initial vaccination through Day 29 visits and subsequent database lock)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Monovalent GI.1 (Experimental): Monovalent GI.1 tableted vaccine group
  Interventions: Biological: VXA-G1.1-NN; Biological: Placebo Tablets
- Monovalent GII.4 (Experimental): Monovalent GII.4 tableted vaccine group
  Interventions: Biological: VXA-G2.4-NS; Biological: Placebo Tablets
- Bivalent GI.1 and GII.4 vaccine group (Experimental): Bivalent vaccine group consisting of co-administration of GI.1 and GII.4 vaccine
  Interventions: Biological: VXA-G1.1-NN; Biological: VXA-G2.4-NS
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Biological: Placebo Tablets

INTERVENTIONS:
Biological: VXA-G1.1-NN — Monovalent GI.1 tableted vaccine
  Other Names: GI.1 oral vaccine tablet
  Arms: Bivalent GI.1 and GII.4 vaccine group; Monovalent GI.1
Biological: VXA-G2.4-NS — Monovalent GII.4 tableted vaccine
  Other Names: GII.4 oral vaccine tablet
  Arms: Bivalent GI.1 and GII.4 vaccine group; Monovalent GII.4
Biological: Placebo Tablets — Tablets matching in number and appearance to active vaccine doses
  Other Names: Oral tablets for control arm
  Arms: Monovalent GI.1; Monovalent GII.4; Placebo

SUMMARY:
VXA-NVV-103 is a phase 1B Randomized, Double-Blind, Placebo-Controlled, Multi-Center Safety and Immunogenicity Study of Adenoviral-vector Based Oral Norovirus Vaccines Expressing GI.1 or GII.4 VP1 with Monovalent or Bivalent Dosing in Healthy Adult Volunteers. The study consists of 2 parts: Part 1 is the double-blinded portion where subjects will be randomized to one of two monovalent vaccine groups, bivalent vaccine group or placebo. Subjects will be followed for ~4 weeks post vaccination for safety and immunogenicity. Part 2 will consist of an open label booster vaccination for the bivalent treatment group ~4 months post initial vaccination. All subjects will be followed for long term safety for 1 year post initial vaccination.

DETAILED DESCRIPTION:
VXA-NVV-103 is a phase 1B Randomized, Double-Blind, Placebo-Controlled, Multi-Center Safety and Immunogenicity Study of Adenoviral-vector Based Oral Norovirus Vaccines Expressing GI.1 or GII.4 VP1 with Monovalent or Bivalent Dosing in Healthy Adult Volunteers. The study consists of 2 parts with will enroll 86 subjects:

Part 1 - Double Blind Period: Post confirmation of eligibility subjects will be randomized in a double-blinded manner to one of four treatment arms. Treatment Group 1 will contain an open-label sentinel group of 6 subjects to be enrolled prior to initiation of subsequent treatment groups. After review of the safety data and confirmation the dose is well tolerated through Study Day 8, the rest of the study will proceed in a double-blinded, randomized fashion. The 6 sentinel subjects will not be part of the 16 subjects in Treatment Group 1 to be enrolled in the double-blinded placebo-controlled cohort; randomization will be 1:1:2:1 for Treatment Groups 1 through 4 respectively.

Study Design and Vaccine Groups

1. Monovalent GII.4 VXA-G2.4-NS (6 sentinels / 16 randomized)
2. Monovalent GI.1 VXA-G1.1-NN (16 randomized)
3. Bivalent GII.4/GI.1 VXA-G2.4-NS + VXA-G1.1-NN (32 randomized)
4. Placebo Tablets no vaccine (16 randomized)

Subjects will be followed for ~4 weeks post vaccination for safety and immunogenicity. The study database will be locked post completion of Day 29 visits.

Part 2 will consist of an open label booster vaccination for the bivalent treatment group ~4 months post initial vaccination. Subjects will be followed for safety and immunogenicity for ~4 weeks post the boost.

All subjects will be followed for long term safety for 1 year post initial vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 to 49 years, inclusive
* General good health, without significant medical illness, based on medical history, physical examination, vital signs, and clinical laboratories
* Demonstrate comprehension of the protocol procedures and willingness to adhere to all visits and assessments
* Body mass index between 17 and 35 at screening
* Female subjects must have a negative pregnancy test at screening and before each vaccination and fulfill protocol specified criteria for adequate birth control.

Exclusion Criteria:

* Presence of a significant medical condition which in the opinion of the investigator precludes participation in the study
* History of cancer or cancer treatment within past 3 years
* Presence of immunosuppression or medical condition possibly associated with impaired immune responsiveness, including diabetes mellitus or angioedema
* Donation or use of blood/blood products within 4 weeks prior to vaccination
* Diagnosed bleeding disorder or significant bruising or bleeding difficulties that could make blood draws problematic.
* Any condition that resulted in the absence or removal of the spleen
* Positive HIV, HBsAg or HCV tests at the screening visit
* Use of antibiotics, proton pump inhibitors, H2 blockers or antacids within 7 days of vaccination
* Use of medications known to affect the immune function within 14 days of vaccination
* Use of NSAIDs, sulfonylureas, and angiotensin II blockers within 7 days of vaccination
* Evidence of recent or of current nonbacterial gastroenteritis suggestive of NV infection to any gastroenteritis within 2 weeks of vaccination
* History of drug, alcohol or chemical abuse within 1 year of screening or positive urine drug test at screening
* Consistent/habitual smoking within 2 months as per medical history
* History of hypersensitivity or allergic reaction to any component of the investigational vaccine or placebo
* Use of any investigational vaccine, drug or device within 8 weeks preceding vaccination, or planned use of the above stated for the duration of the study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Rate of Solicited Adverse Events | Day 1 (Vaccination) to 7 days post vaccination
  Comparison of rate of occurance and severity of Solicited Adverse Events observed between treatment groups
Rate of Unsolicited Adverse Events | Day 1 (Vaccination) to 28 days post vaccination
  Comparison of the rate of occurrence and severity of unsolicited Adverse Events observed between treatment groups
Immunogenicity - VP1 Specific IgA ASC | Day 1 (vaccination) to 7 days post-vaccination
  LS Mean difference in VP1 specific IgA ASC between vaccine and placebo group
Immunogenicity - BT50 Assay | Day 1 (vaccination) to 28 days post-vaccination
  Difference in HBGA blocking antibodies (by blocking titer fifty assay [BT50]) between vaccine and placebo groups

SECONDARY OUTCOMES:
Immunogenicity - VP1 specific serum IgG | Day 1 (vaccination) to 7 days post-vaccination
  LS Mean difference in VP1 specific serum IgG between vaccine and placebo groups

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Manning, MD, Principal Investigator — Rapid Medical Research
Locations (1):
- Rapid Medical Research, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Study results will be summarized and presented by treatment arm comparisons. Individual subject data will not be shared with other researchers.